CLINICAL TRIAL: NCT07279610
Title: N-Acetylcysteine as Therapy for Transplantation- Associated Thrombotic Microangiopathy
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOOCHOW-HY-2024
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-02

CONDITIONS: Thrombotic Microangiopathy
MeSH Terms: conditions — Thrombotic Microangiopathies | interventions — Acetylcysteine; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NAC (Experimental): N-acetylcysteine injection will be administered intravenously to TA-TMA patients at a total daily dose of 16g. The daily dose is divided into two equal doses of 8g each, administered in the morning and evening. Each 8g dose is to be infused over a period of 1 hour. This regimen continues for 14 consecutive days.
  Interventions: Drug: N-Acetylcysteine (NAC) Treatment

INTERVENTIONS:
Drug: N-Acetylcysteine (NAC) Treatment — N-acetylcysteine injection will be administered intravenously to TA-TMA patients at a total daily dose of 16g. The daily dose is divided into two equal doses of 8g each, administered in the morning and evening. Each 8g dose is to be infused over a period of 1 hour. This regimen continues for 14 consecutive days.

SUMMARY:
This multicenter, prospective, single-arm clinical trial aims to evaluate the efficacy and safety of N-acetylcysteine (NAC) for treating Transplantation-Associated Thrombotic Microangiopathy (TA-TMA), a severe complication of hematopoietic stem cell transplantation characterized by microangiopathic hemolytic anemia, thrombocytopenia, and organ injury, with an incidence of 4%-30%. Current treatments, including plasma exchange (response rate <10%) and costly complement inhibitors like Eculizumab (71% response) which are not widely accessible, are inadequate. Inspired by NAC's success in treating the related condition thrombotic thrombocytopenic purpura (TTP) and supported by bioinformatic analyses of patient data revealing enhanced oxidative stress pathways and identifying NAC as a potential targeted therapy, our prior study demonstrated that NAC prophylaxis significantly reduces TA-TMA incidence and improves survival. Building on this promising foundation, this study will enroll patients meeting TA-TMA diagnostic criteria for NAC treatment, assessing its potential as a safe, effective, and affordable therapeutic option.

DETAILED DESCRIPTION:
Background:

Transplantation-associated thrombotic microangiopathy (TA-TMA) is a severe complication of hematopoietic stem cell transplantation, characterized by microangiopathic hemolytic anemia, thrombocytopenia, elevated lactate dehydrogenase, elevated serum creatinine, schistocytes on peripheral blood smear, and microvascular thrombosis. Its pathogenesis is associated with complement system activation leading to endothelial injury. The incidence of TA-TMA ranges from 4% to 30%. Current treatments, including withdrawal of calcineurin inhibitors, switching to other immunosuppressants, and plasma exchange (which has a response rate below 10%), are unsatisfactory. Complement-targeted therapies like the C5 monoclonal antibody Eculizumab and the lectin pathway inhibitor Narsoplimab show promise with response rates of 71% and 61%, respectively. However, their high cost and limited availability (e.g., some are not accessible in China) restrict widespread use. There is a clear lack of prospective clinical trials for TA-TMA treatment.

Thrombotic thrombocytopenic purpura (TTP) shares similar clinical features with TA-TMA. In 2016, N-acetylcysteine (NAC) combined with plasma exchange achieved complete remission in three refractory TTP patients. NAC, a safe, economical, and readily available antioxidant, is approved for acetaminophen toxicity and COPD. It inhibits platelet adhesion to von Willebrand factor (VWF) by reducing disulfide bonds in VWF, thereby decreasing the size of soluble high molecular weight VWF multimers, as validated in animal TTP models. This success in TTP suggests a potential therapeutic direction for TA-TMA.

Analysis of RNA sequencing data from TA-TMA patients in the GEO database revealed enhanced oxidative stress-related gene expression. Furthermore, whole-genome sequencing of a TA-TMA patient's blood and analysis via the IPA database identified NAC as a potential effective treatment. A subsequent prospective trial demonstrated that NAC prophylaxis significantly reduced TA-TMA incidence, delayed its onset, and improved event-free survival in transplant patients. However, no clinical trial has yet investigated NAC for the treatment of established TA-TMA. Compared to expensive complement inhibitors, NAC represents a safe, accessible, and affordable drug with the potential to offer effective and feasible therapy for TA-TMA patients.

Objective:

To evaluate the efficacy and safety of N-acetylcysteine in patients with diagnosed TA-TMA.

Study Design:

This is a multicenter, prospective, single-arm clinical study.

Methods:

Patients who meet the TA-TMA diagnostic criteria will be screened based on predefined inclusion and exclusion criteria. Enrolled patients will receive N-acetylcysteine treatment. The primary endpoints will be the assessment of treatment efficacy (including response rates) and safety (monitoring of adverse events).

ELIGIBILITY:
Inclusion Criteria:

- 1. Informed Consent: The patient must have the ability to understand and the willingness to participate in the study and must sign a written Informed Consent Form.

2. Age: ≥ 18 years old, regardless of gender. 3. Diagnosis: Subjects diagnosed with TA-TMA according to the Harmonizing Definitions, defined as meeting one of the following:

* TA-TMA confirmed by renal or intestinal biopsy, OR
* Fulfilling at least four of the following seven clinical or laboratory criteria within a 14-day period:

  1. Anemia, defined as persistent transfusion dependence after myeloid engraftment, OR a decrease in hemoglobin >10 g/L, OR new-onset transfusion dependence.
  2. Thrombocytopenia, defined as failure of platelet engraftment, OR a higher-than-expected platelet transfusion requirement, OR refractory platelet transfusion, OR a >50% decrease in platelets after initial engraftment.
  3. Lactate dehydrogenase (LDH) level above the upper limit of normal (ULN).
  4. Presence of schistocytes on peripheral blood smear.
  5. Hypertension (blood pressure ≥140/90 mmHg).
  6. sC5b-9 level above the ULN.
  7. Proteinuria (random urine protein-to-creatinine ratio ≥1 mg/mg).

     Exclusion Criteria:
     * 1. The subject has received complement blockade therapy (e.g., Eculizumab or Narsoplimab) within the past 3 months.

       2. The subject has a history of drug and/or alcohol abuse within the 6 months prior to enrollment.

       3. The subject has a life expectancy of less than 3 months. 4. The subject is considered by the investigator to be unable or unwilling to cooperate with the study procedures.

       5. The subject is a family member or employee of the investigator. 6. The patient is pregnant or lactating. 7. The subject has a history of Human Immunodeficiency Virus (HIV) infection. 8. The subject has a known allergy to any component of the investigational drug (N-acetylcysteine).

       9. The subject has cardiac insufficiency, defined as an ejection fraction (EF) <30%, or NYHA Class III or higher heart failure, or other cardiac conditions deemed by the investigator as unsuitable for enrollment.

       10. The subject has contraindications to N-acetylcysteine, such as active bronchial asthma or peptic ulcer disease.

       11. The patient refuses to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The efficacy of N-acetylcysteine treatment for TA-TMA | Day 1 to 60 days after the enrollment of N-acetylcysteine
  Evaluate the efficacy of N-acetylcysteine in patients with TA-TMA by response defined as:
  1. Improvement in TMA laboratory markers of platelet count and lactate dehydrogenase (LDH), and
  2. Improvement in clinical status

SECONDARY OUTCOMES:
100-day survival | Study Day of TA-TMA diagnosis to 100 days later
  Number of participants alive from the date of TMA diagnosis
Platelet count change from baseline | Study Day 1 to Day 60
  Changes from baseline in Platelet count
Change From Baseline in LDH | Study Day 1 to Day 60
  Changes from baseline in LDH
Change From Baseline in Hemoglobin | Study Day 1 to Day 60
  Change From Baseline in Hemoglobin
Change From Baseline in Creatine | Study Day 1 to Day 60
  Change From Baseline in Creatine
Freedom From Platelet Transfusion | Study Day -14 to Day 60 following the last platelet transfusion
  Number of participants with absence of platelet transfusions
Freedom From Red Blood Cell (RBC) Transfusion | Study Day -14 to Day 60 following the last RBC transfusion
  Number of participants with absence of RBC transfusions
Adverse events | 2 years
  Adverse events are evaluated with CTCAE V5.0.
Overall Survival (OS) | 2 years
  Time from enrollment to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pan T, Qi J, Tang Y, Yao Y, Chen J, Wang H, Yang J, Xu X, Shi Q, Liu Y, He X, Chen F, Ma X, Hu X, Wu X, Wu D, Han Y. N-Acetylcysteine as Prophylactic Therapy for Transplantation-Associated Thrombotic Microangiopathy: A Randomized, Placebo-Controlled Trial. Transplant Cell Ther. 2022 Nov;28(11):764.e1-764.e7. doi: 10.1016/j.jtct.2022.07.029. Epub 2022 Aug 5. PMID 35940529
- [Result] Qi J, Hu S, He X, Pan T, Yang L, Zhang R, Tang Y, Wu D, Han Y. N-Acetyl-L-Cysteine Potentially Inhibits Complement Activation in Transplantation-Associated Thrombotic Microangiopathy. Transplant Cell Ther. 2022 Apr;28(4):216.e1-216.e5. doi: 10.1016/j.jtct.2021.12.018. Epub 2021 Dec 31. PMID 34979328
- [Result] Tersteeg C, Roodt J, Van Rensburg WJ, Dekimpe C, Vandeputte N, Pareyn I, Vandenbulcke A, Plaimauer B, Lamprecht S, Deckmyn H, Lopez JA, De Meyer SF, Vanhoorelbeke K. N-acetylcysteine in preclinical mouse and baboon models of thrombotic thrombocytopenic purpura. Blood. 2017 Feb 23;129(8):1030-1038. doi: 10.1182/blood-2016-09-738856. Epub 2016 Dec 23. PMID 28011677
- [Result] Chen J, Reheman A, Gushiken FC, Nolasco L, Fu X, Moake JL, Ni H, Lopez JA. N-acetylcysteine reduces the size and activity of von Willebrand factor in human plasma and mice. J Clin Invest. 2011 Feb;121(2):593-603. doi: 10.1172/JCI41062. Epub 2011 Jan 25. PMID 21266777
- [Result] Zhang R, Zhou M, Qi J, Miao W, Zhang Z, Wu D, Han Y. Efficacy and Safety of Eculizumab in the Treatment of Transplant-Associated Thrombotic Microangiopathy: A Systematic Review and Meta-Analysis. Front Immunol. 2021 Jan 20;11:564647. doi: 10.3389/fimmu.2020.564647. eCollection 2020. PMID 33552043
- [Result] Schoettler ML, Carreras E, Cho B, Dandoy CE, Ho VT, Jodele S, Moissev I, Sanchez-Ortega I, Srivastava A, Atsuta Y, Carpenter P, Koreth J, Kroger N, Ljungman P, Page K, Popat U, Shaw BE, Sureda A, Soiffer R, Vasu S. Harmonizing Definitions for Diagnostic Criteria and Prognostic Assessment of Transplantation-Associated Thrombotic Microangiopathy: A Report on Behalf of the European Society for Blood and Marrow Transplantation, American Society for Transplantation and Cellular Therapy, Asia-Pacific Blood and Marrow Transplantation Group, and Center for International Blood and Marrow Transplant Research. Transplant Cell Ther. 2023 Mar;29(3):151-163. doi: 10.1016/j.jtct.2022.11.015. Epub 2022 Nov 25. PMID 36442770

DOCUMENTS (1):
  • Informed Consent Form (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT07279610/ICF_000.pdf